CLINICAL TRIAL: NCT04036032
Title: Role of Aerobic Exercise to Modulate Cardiotoxicity in Long Term Cancer Survivors Exposed to Anthracycline Therapy
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tiffany Ruiz, Cardio-oncology nurse program manager, Connecticut Children's Medical Center
Other Study IDs: 14-110
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Cardiotoxicity
MeSH Terms: conditions — Neoplasms; Cardiotoxicity | interventions — Resistance Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens collected for micro RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise program — Encourage to work out 4 to 5 times a week for 3 months. Patient chooses what exercise they would like to do. At YMCA visit for fitness assessments they provide exercise support

SUMMARY:
Over 50% of the more than 270,000 childhood cancer survivors in the U.S. have been treated with anthracyclines and thus are at risk of developing cardiotoxicity. The impact of exercise training on LV structure has been extensively studied. Left ventricular hypertrophy and cardiac chamber enlargement with the accompanying ability to generate a large stroke volume are direct results of exercise training. Aerobic exercise therapy offers a non-pharmacological mechanism to modulate multiple gene expression pathways that may promote cardiac remodeling. No prior studies have investigated the efficacy of aerobic exercise in the prevention or treatment of anthracycline-induced cardiotoxicity. We hypothesize that exercise intervention leads to a reverse in adverse cardiac remodeling with improvement of global and regional myocardial function in patients exposed to anthracycline.

DETAILED DESCRIPTION:
The goal of this research is to assess the effect of exercise intervention on imaging parameters by CMR, cardiopulmonary indices and MicroRNA expression in survivors of childhood cancer exposed to anthracycline therapy. Thus, results from this study could provide a foundation for a paradigm shift in our approach to the prevention and management of anthracycline induced cardiotoxicity in this population. Patients who have been exposed to anthracycline treatment and who are greater than 9 years of age will be enrolled.

Patients will come into the clinic for 7 study visits. Patients will have an exercise intervention provided to them by a trainer at the designated YMCA. Patients will start their exercise for 15 minutes per day for 3-5 days a week for week one progressing to 45 minutes per day, 3 - 5 days a week as tolerated by the end of week four. The goal during each session is for the patient to exercise at 50-80% of their age adjusted maximum heart rate, which will be determined by the personal trainer (PT) at their initial visit. The exercise program will continue for 12 weeks (ending at 16 weeks after entry to the study).

In the clinic patients will have the following tests completed:

Week 0 and Week 16: Cardiac MRI, stress test along with blood samples and Karnofsky/Lansky Scale.

Week 0 patients receive a Fitbit and home diary/Wellness Log for completion. Week 4 began exercise intervention Weeks 0, 4, 8, 16 and 20 patients will receive phone calls for symptom tracker Weeks 0, 16, and 6 month f/u patients complete a questionnaire

Patients will also have Fitness assessments to see how their exercise intervention is doing.

Specific Aim 1: To measure the impact of the toolbox exercise intervention on cardiac remodeling as measured by cardiac magnetic resonance Imaging (CMR) in childhood cancer survivors exposed to Anthracycline therapy. The objective of this Aim is to use CMR to characterize changes of myocardial mass, volume, global and regional myocardial function at baseline and following exercise intervention.

Specific Aim 2a: To examine the impact of the toolbox exercise intervention on exercise testing derived cardiopulmonary parameters in childhood cancer survivors exposed to Anthracycline therapy. The objective of this aim is to assess changes in oxygen consumption (peak VO2), VO2 @ anaerobic threshold, O2 pulse, and he ventilation/carbon dioxide slope (VE/VCO2slope) at baseline and following exercise intervention.

Specific Aim 2b: To examine the impact of the toolbox exercise intervention on quality of life, functional status and fitness in childhood cancer survivors exposed to anthracycline therapy. his Aim will test the hypothesis that exercise intervention will result in improvement in:

1. Quality of life as measured by PedsQL 4.0 for children ≤ 18 and the SF-36 for adults > 18
2. Patient functional status as measured by the Karnofsky/Lansky Scale
3. Fitness as measured by range of motion, balance, endurance, body composition and and functional strength

Specific Aim 3: Analyze serum microRNA (miRNA) expression focusing on cardiac stress signaling pathways at three time points during each stress test: at baseline (prior to stress testing), immediately post-exercise (within 1min of completion of exercise testing), and after 1 hour of rest following stress testing). The objective of this aim is to measure changes in microRNA expression in plasma related to stress signaling pathways after exercise intervention when compared to baseline

ELIGIBILITY:
Inclusion Criteria:

* Long-term childhood cancer survivors greater than 9 years of age*
* Exposed to anthracycline chemotherapy * Age > 9 years of age was chosen to avoid the need for general anesthesia or sedation

Exclusion Criteria:

* Contraindications to CMRI*
* Individuals needing sedation to complete the cMRI
* Subject not able to perform stress test.
* Pregnancy**
* Non-English speaking individuals
* Orbital X-Ray confirmed to have metal in the eye or patient confirmed to have metal in the eye

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are over 9 years of age and who have had anthracycline chemotherapy treatments that were completed over 2 years ago will be asked to participant in the study.
  Patients from the oncology clinic and the Stars clinic will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Small increase in the left and right ventricular volume | Baseline to Week 12
  Small increase in the left and right ventricular volume
Small increase in left and right ventricular mass | Baseline to Week 12
  Small increase in left and right ventricular mass

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Berthod (Ruiz), MSN, RN, CPN, CCRC, Principal Investigator — Connecticut Children's Medical Center
Locations (2):
- United States (2):
  - CT Children's Medical Center, Hartford, Connecticut
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Pending information from PI